CLINICAL TRIAL: NCT02608632
Title: High Frequency Guided Renal Artery Denervation for Improving Outcome of Renal Ablation Procedure
Brief Title: HFS-guided Renal Ablation for Improving Outcome of Renal Denervation Procedure
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 7452RDNHFS
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Hypertension
Keywords: Renal denervation; Ablation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (RDN guided by HFS) (Experimental): Renal arteries were assessed for suitability of ablation by renal angiography. The real-time 3-dimensional aorta-renal artery maps were reconstructed with the use of navigation system and ablation catheter via femoral artery access. After that high-frequency stimulation (HFS) was used before the initial and after each radiofrequency (RF) delivery within the renal artery. RDN was considered to have been achieved when the sudden increase of blood pressure (> 15 mm Hg from invasive arterial monitoring) was eliminated in response to HFS.
  RF ablations of 8-12 watts (impedance drop >10%) were applied discretely from the first distal main renal artery bifurcation all the way back to the ostium. The duration of each RF delivery was 60-120 sec, and up to 6 lesions (separated by > 5 mm) were performed both longitudinally and rotationally within each renal artery.
  Interventions: Device: Renal denervation guided by HFS
- Group 2 (RDN as standard procedure) (Active Comparator): Renal arteries were assessed for suitability of ablation by renal angiography. The real-time 3-dimensional aorta-renal artery maps were reconstructed with the use of navigation system and ablation catheter via femoral artery access.
  RF ablations of 8-12 watts (impedance drop >10%) were applied discretely from the first distal main renal artery bifurcation all the way back to the ostium. The duration of each RF delivery was 60-120 sec, and up to 6 lesions (separated by > 5 mm) were performed both longitudinally and rotationally within each renal artery. High-frequency stimulation (HFS) was performed before and after RDN to just to verify the response of BP
  Interventions: Device: Renal denervation as standard procedure

INTERVENTIONS:
Device: Renal denervation guided by HFS
  Arms: Group 1 (RDN guided by HFS)
Device: Renal denervation as standard procedure
  Arms: Group 2 (RDN as standard procedure)

SUMMARY:
To increase the number of responders using HFS-guided renal artery denervation (RDN) in patients with resistant and moderate resistant hypertension

ELIGIBILITY:
Inclusion Criteria:

* Office-based systolic blood pressure of ≥140/90 mm Hg and <160/100 mm Hg (moderate resistant hypertension) or ≥160/100 mm Hg (severe resistant hypertension), despite treatment with 3 antihypertensive drugs (including a diuretic).
* A glomerular filtration rate ≥45 mL/min/1⋅73 m2, with modification of diet using a renal disease formula.

Exclusion Criteria:

* Secondary causes of hypertension
* Severe renal artery stenosis or dual renal arteries
* Congestive heart failure
* Left ventricular ejection fraction <35%
* Previous renal artery stenting or angioplasty
* Type 1 diabetes mellitus

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-12 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
number of responders to renal denervation procedure | 12 month

SECONDARY OUTCOMES:
complications rate | 12 month
cross-over rate | 12 month

CONTACTS AND LOCATIONS:
Locations (3):
- Russia (3):
  - Federal Center of Cardiovascular surgery, Krasnoyarsk
  - Regional Hospital, Krasnoyarsk
  - Federal Center of Prophylactic Medicine, Moscow